CLINICAL TRIAL: NCT06373562
Title: The Influence of Sports and Hypoxic Training on the Regeneration and Adaptation of Skeletal Muscles to Exercise in Wrestlers.
Brief Title: Effect of Hypoxic Exposure on Blood Variables in Elite Wrestlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Wrestlers LH-TL
Record Dates: First submitted 2024-04-12; First posted 2024-04-18 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-04

CONDITIONS: Hypoxia
Keywords: hypoxia; EPO; wrestlers; HIF-1; athletes
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Wrestlers in H group were living in hypoxic rooms for 8-14h/d and between that they were participating in sports training. C group was participating in the same training protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxia (Experimental): Live High-Train Low method was used.
  Interventions: Other: hypoxia
- Control group (No Intervention): The control group was participating in the same training protocol.

INTERVENTIONS:
Other: hypoxia — The athletes were living in hypoxic rooms, which could simulate a selected altitude above sea level.
  Arms: Hypoxia

SUMMARY:
Twelve male wrestlers of the National Polish Team were observed in the study during the camp. The hypoxia group (n=6) participated in sports training and hypoxic exposure, while the control group (n=6) included wrestlers participating only in sports training. The hypoxic group lived and slept in hypoxic rooms. During the camp, all wrestlers followed the same training schedule and diet. In the blood were determined levels of creatine kinase (CK), C-reactive protein (hsCRP) concentration, nitric oxide (NO), morphology, reticulocytes, lipid profile, and ferritin. Also vascular endothelial growth factor (VEGF, VEGFR2, and VEGFR3), erythropoietin (EPO), angiopoietin (Ang 1, Ang 2), endothelial cell adhesion factor-1 (VCAM-1), Erythropoietin (EPO) and hypoxia-inducible factor 1 (HIF-1). Body weight composition was determined.

DETAILED DESCRIPTION:
Hypoxia exposure applied to professional athletes has attracted attention and scientific debate due to its effects on improving physiological response through cardiovascular and hematological mechanisms. Presently, hypoxic training programs are developed to improve exercise performance in athletes, a useful training method for athletes that may improve their performance in future sea-level competitions. 12 males were divided into the hypoxic (H) and control (C) groups. Group H was living and sleeping in hypoxic rooms (method live high-train low) for 8-14h/d (FiO2≈14%). The implementation of the project was intended to: 1) assess the dynamics of changes in the concentration of pro-inflammatory indicators and hematopoiesis in athletes to variable training loads and hypoxia, 2) explain the usefulness of hypoxic exposure in adaptation to physical exercise, 3) observe the length of the hypoxic cycle necessary to maintain the effect of high-altitude training. In the blood serum the level of basic biochemical indicators of fatigue related to muscle damage, inflammation, and energy deficit, i.e. total creatine kinase (CK) activity, C-reactive protein (hsCRP) concentration, nitric oxide (NO). Moreover, basic hematological indicators: morphology, reticulocytes, lipid profile, and ferritin. Also, angiogenesis regulators: vascular endothelial growth factor (VEGF) and VEGF receptors (VEGFR2 and VEGFR3), erythropoietin (EPO), angiopoietin (Ang 1, Ang 2), endothelial cell adhesion factor-1 (VCAM-1), Erythropoietin (EPO) and hypoxia-inducible factor 1 (HIF-1). Body weight composition was determined using a body analyzer. Further investigations into hypoxia methods while considering individual capabilities are necessary for gaining deeper insights, into how hypoxia affects blood count and different blood variables among athletes.

ELIGIBILITY:
Inclusion Criteria:

* member of national wrestler's teams, and sports camp participant.

Exclusion Criteria:

* negative symptoms of hypoxia, and/or injury.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2013-12-18 (Actual); Study Completion 2013-12-18 (Actual)

PRIMARY OUTCOMES:
CK | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  creatine kinase
hsCRP | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  reactive C-protein
HIF-1 | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  hypoxia-inducible factor 1
EPO | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  Erythropoietin
VEGF, VEGF 2, VEGF 3. | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  vascular endothelial growth factor
Ang 1, Ang 2 | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  angiopoietin
VCAM-1 | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  endothelial cell adhesion factor-1

OTHER OUTCOMES:
blood count | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  morphology
lipid profile | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  HDL, LDL, triglycerides
ferritin | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  ferritin
(untitled outcome) | The blood was taken at the beginning of the camp (baseline), after 6 days, after 15 days.
  nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kasperska, Principal Investigator — Poznań University of Physical Education, Faculty of Sport Sciences in Gorzów Wielkopolski, Poland;

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasperska A, Zembron-Lacny A. The effect of intermittent hypoxic exposure on erythropoietic response and hematological variables in elite athletes. Physiol Res. 2020 Apr 30;69(2):283-290. doi: 10.33549/physiolres.934316. Epub 2020 Mar 23. PMID 32199016
- [Background] Czuba M, Fidos-Czuba O, Ploszczyca K, Zajac A, Langfort J. Comparison of the effect of intermittent hypoxic training vs. the live high, train low strategy on aerobic capacity and sports performance in cyclists in normoxia. Biol Sport. 2018 Mar;35(1):39-48. doi: 10.5114/biolsport.2018.70750. Epub 2017 Oct 11. PMID 30237660
- [Background] Wilber RL. Application of altitude/hypoxic training by elite athletes. Med Sci Sports Exerc. 2007 Sep;39(9):1610-24. doi: 10.1249/mss.0b013e3180de49e6. PMID 17805095
- [Background] Li J, Li Y, Atakan MM, Kuang J, Hu Y, Bishop DJ, Yan X. The Molecular Adaptive Responses of Skeletal Muscle to High-Intensity Exercise/Training and Hypoxia. Antioxidants (Basel). 2020 Jul 24;9(8):656. doi: 10.3390/antiox9080656. PMID 32722013